CLINICAL TRIAL: NCT04186741
Title: Inner and Middle Ear Effects of Hyperbaric Oxygen Therapy
Brief Title: Inner and Middle Ear Effects of Hyperbaric Oxygen Thrapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nahla Ahmed Abd elhafez Mousa, Principle investigator, Assiut University
Other Study IDs: IMO
Record Dates: First submitted 2019-11-15; First posted 2019-12-05 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2019-12

CONDITIONS: Otitic Barotrauma
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HBO Group: Patients already recieving hyperbaric oxygen therapy for treatment of other medical conditions requiring it as in diabetic foot , cerebral infarctions
  Interventions: Drug: Hyperbaric oxygen

INTERVENTIONS:
Drug: Hyperbaric oxygen — Patients already on treatment by hyperbaric oxygen therapy for medical conditions requiring treatment by it

SUMMARY:
Audiological evaluation performed to patients on hyperbaric oxygen therapy to see its effects on middle ear pressure

DETAILED DESCRIPTION:
Thirty patients will be recruited from center pf hyperbaric oxygen therapy Every patient who received HBOT was submitted for Demographic data:age,gender,condition raquiring HBOT,use of analgesics,history of diabets ,cardiovascular or respiratory disease ,psychatric illness,smoking history facial/ENT problems and previous HBOT problems then tympanometry and basic pure tone audiometry including air and bone conduction is done following each of the first five treatment

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years old already recieving hyperbaric oxygen therapy for treatment of other medical conditions required treatment by it as in diabetic foot

Exclusion Criteria:

* patients who already had tympanostomy tubes

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Measument of middle ear pressure after exposure to hyper baric oxygen therapy
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Changing in middle ear pressure | Through completion of study after 2 years
  Measuring middle ear pressure before exposure ro hyperbaric oxygen and following each of the first five treatments

CONTACTS AND LOCATIONS:
Overall Officials: Enas S Mohamed, Professor, Principal Investigator — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Result] Yamamoto Y, Noguchi Y, Enomoto M, Yagishita K, Kitamura K. Otological complications associated with hyperbaric oxygen therapy. Eur Arch Otorhinolaryngol. 2016 Sep;273(9):2487-93. doi: 10.1007/s00405-015-3845-9. Epub 2015 Dec 9. PMID 26650550